CLINICAL TRIAL: NCT04020874
Title: Reducing Head Impact Exposure in Hawaiian Football Players and Enhancing Community Awareness and Environment for Head-Safety
Brief Title: Reducing Head Impact Exposure in Hawaii High School Football
Acronym: HuTT808
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: Gary O. Galiher Foundation (Unknown); University of Hawaii (Other); University of Michigan (Other); Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Erik Swartz, Professor and Department Chair, University of Massachusetts, Lowell
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HuTT808
Record Dates: First submitted 2019-07-01; First posted 2019-07-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Head Trauma; Cognitive Change; Confidence, Self; Sports Injuries in Children
Keywords: concussion; tackle; youth sports
MeSH Terms: conditions — Craniocerebral Trauma; Brain Concussion

STUDY DESIGN:
Intervention Model Description: pre-test, post-test, quasi-experimental
Who Masked: Investigator
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): Year 1, no intervention to generate baseline, comparative data for subsequent years
- HuTT-2x (Experimental): The HuTT® program emphasizes proper tackling and blocking techniques using a progressive series of closely supervised drills. Skill rehearsal is done without helmets and shoulder pads and is the inherent element of HuTT® in order to reinforce behaviors which remove the head as a point of contact. The HuTT® program is modeled after basic tackling/blocking drills familiar to the sport of football. Feedback to confirm or correct proper skill development is provided by coaches trained in the HuTT® technique. HuTT® drills are conducted at an intensity of 50-75% effort and over a period of approximately 10 minutes. The intervention will be conducted 2 times each week throughout the regular season.
  Interventions: Behavioral: HuTT-2x
- HuTT-4x (Experimental): The HuTT® program emphasizes proper tackling and blocking techniques using a progressive series of closely supervised drills. Skill rehearsal is done without helmets and shoulder pads and is the inherent element of HuTT® in order to reinforce behaviors which remove the head as a point of contact. The HuTT® program is modeled after basic tackling/blocking drills familiar to the sport of football. Feedback to confirm or correct proper skill development is provided by coaches trained in the HuTT® technique. HuTT® drills are conducted at an intensity of 50-75% effort and over a period of approximately 10 minutes. The intervention will be conducted 4 times each week throughout the regular season.
  Interventions: Behavioral: HuTT-4x

INTERVENTIONS:
Behavioral: HuTT-2x — tackling and blocking training twice/week
  Arms: HuTT-2x
Behavioral: HuTT-4x — tackling and blocking training four times/week
  Arms: HuTT-4x

SUMMARY:
This three-year study will determine the effectiveness of a helmetless tackling training intervention to decrease head impact exposure in Hawaiian high school football players.

DETAILED DESCRIPTION:
High school football participants are reported to sustain an average of 600, and as many as 2000, head impacts in a single season. Impacts to the top and front of the helmet generate the greatest forces, and thus pose the highest risk for acute brain and spinal cord injury. Equally disconcerting is the potential relationship between the accumulation of concussive and sub-concussive impacts (head impact exposure, HIE) and the risk for developing long-term conditions such as cognitive impairment, early-onset Alzheimer's, and chronic traumatic encephalopathy (CTE). Tackling and blocking behaviors using the head as the point of first contact can be attributed, in part, to the fact that players wear a helmet, which influences behavior by increasing the perception of safety.

The central hypothesis is such that a football player who regularly practices tackling and blocking drills without a helmet in a controlled environment will naturally leave the head out of contact and is likely to continue to do so while wearing the helmet during games and full-contact practices. This learned motor behavior will reduce the number of head impacts a football player experiences throughout their playing career and thus reduces the risk of acute and chronic head and neck injury.

The investigation will be a pre-test, post-test quasi experimental design using an evidence-based helmetless tackling and blocking program (HuTT®) with football players (~200) recruited from high school football teams in Oahu, Hawaii.

Year 1 will serve as a baseline and entail collecting only head impact data during regular football participation for two teams. After adding a third team for years 2 and 3, all subjects will then undergo the HuTT® Program intervention emphasizing proper tackling and blocking techniques under closely supervised drills where players participate without their helmets and shoulder pads in place.

From the outset, subjects will use a new Speedflex helmet outfitted with the InSite™ head impact sensor (Riddell, Co). The helmet and sensor will be worn in all practices and games and used to record head impact exposure (frequency, location, and magnitude). ImPACT tests will be conducted at pre- and post-season intervals to measure verbal and visual memory composite, visual motor speed composite, reaction time composite and symptoms scores. In addition, player self-efficacy for head-safe behavior will be scored each year using a self-reported survey.

A between-subjects ANOVAs will be used to compare outcome measures among teams. Significant interactions and main effects will be identified by appropriate t-tests with Bonferonni corrections at an alpha-level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* be a member on one (junior varsity or varsity) of the participant schools' interscholastic football teams

Exclusion Criteria:

* none

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 496 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Head Impact Exposure Change from Baseline | At the end of three (3) regular football seasons. Season 1 as baseline, seasons 2 and 3 compared against season 1. Each season spanning approximately 13 weeks (July - October)
  The number, force, and location of impacts to the head/helmet of a participant during practices and games as measured by InSite (Riddell)
Neurocognitive performance Change from Baseline | Before and at the end of three (3) regular football seasons. Season 1 as baseline, seasons 2 and 3 compared against season 1. Each season spanning approximately 13 weeks (July - October)
  Pre- and post-season neurocognitive scores (composite values for visual memory, verbal memory, reaction time, visual motor speed)
Self-report Symptom Scores Change from Baseline | At the end of three (3) regular football seasons. Season 1 as baseline, seasons 2 and 3 compared against season 1. Each season spanning approximately 13 weeks (July - October)
  Concussion symptom scores (0-6 Likert scale; 0=none, 1=mild, 6=severe) for 22 symptoms as measured by Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT). Scores are totaled.
Player self-efficacy for achieving and reinforcing head protective behaviors during tackling and blocking Change from Baseline | At the end of three (3) regular football seasons. Season 1 as baseline, seasons 2 and 3 compared against season 1. Each season spanning approximately 13 weeks (July - October)
  Self-efficacy scores on a scale of 0-10 (0=not confident; 10=highly confident) as measured by self-reported tackling and blocking appraisal inventory.
Coach self-efficacy for achieving and reinforcing head protective behaviors during tackling and blocking Change from Baseline | At the end of three (3) regular football seasons. Season 1 as baseline, seasons 2 and 3 compared against season 1.Each season spanning approximately 13 weeks (July - October)
  Self-efficacy scores on a scale of 0-10 (0=not confident; 10=highly confident) as measured by self-reported tackling and blocking appraisal inventory.

SECONDARY OUTCOMES:
Intervention frequency (ie. dose response) | During two (2) regular football seasons. Each season spanning approximately 13 weeks (July - October)
  Dose response effect as measured by head impact exposure

CONTACTS AND LOCATIONS:
Overall Officials: Erik Swartz, Principal Investigator — University of Massachussetts Lowell
Locations (1):
- University of Hawaii at Manoa, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be made available to other researchers